CLINICAL TRIAL: NCT00064181
Title: Irinotecan Combined With Infusional 5-FU/Folinic Acid or Capecitabine and the Role of Celecoxib in Patients With Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy With or Without Celecoxib in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: EORTC-40015; EORTC-40015
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Celecoxib; Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: capecitabine
Drug: celecoxib
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as irinotecan, capecitabine, leucovorin, and fluorouracil use different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of colorectal cancer by stopping blood flow to the tumor. It is not yet known which combination chemotherapy regimen with or without celecoxib is more effective in treating metastatic colorectal cancer.

PURPOSE: This randomized phase III trial is studying two combination chemotherapy regimens and celecoxib to see how well they work compared to two combination chemotherapy regimens alone in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free survival of patients with metastatic colorectal cancer treated with capecitabine and irinotecan vs fluorouracil, leucovorin calcium, and irinotecan with vs without celecoxib.
* Compare the safety of these regimens in these patients.
* Compare the response rate in patients treated with these regimens.
* Compare the time to treatment failure and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind*, multicenter study. Patients are stratified according to participating center, prior adjuvant therapy (yes vs no), and risk group (poor vs intermediate vs good). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive irinotecan IV over 30-90 minutes on days 1 and 22; oral capecitabine twice daily on days 1-15 and 22-36; and oral celecoxib twice daily on days 1-42.
* Arm II: Patients receive irinotecan and capecitabine as in arm I and oral placebo twice daily on days 1-42.
* Arm III: Patients receive irinotecan IV over 30-90 minutes on days 1, 15, and 29; leucovorin calcium (CF) IV over 2 hours and fluorouracil (5-FU) IV over 22 hours on days 1, 2, 15, 16, 29, and 30; and oral celecoxib twice daily on days 1-42.
* Arm IV: Patients receive irinotecan, CF, and 5-FU as in arm III and oral placebo twice daily on days 1-42.

In all arms, treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. If all chemotherapy is discontinued due to toxicity, patients may continue celecoxib or placebo until disease progression, unacceptable toxicity, or starting a new cytotoxic regimen.

NOTE: *The double-blind treatment only applies to the celecoxib and placebo randomization

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 692 patients (173 per treatment arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum
* Metastatic disease
* Measurable disease

  * Patients who received prior radiotherapy must have measurable or evaluable disease outside the radiotherapy field
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN (5 times ULN in the presence of liver metastases)

Renal

* Creatinine clearance at least 51 mL/min
* No severe renal impairment

Cardiovascular

* No severe cardiac disease
* No uncontrolled angina pectoris
* No myocardial infarction within the past 6 months

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study participation
* No active Crohn's disease
* No other malignancy except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No other uncontrolled severe medical condition
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent active or passive immunotherapy for colon cancer

Chemotherapy

* No prior chemotherapy for metastatic disease

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 6 months since prior adjuvant therapy
* More than 4 weeks since prior investigational drugs
* No concurrent sorivudine or chemically related analogues (e.g., brivudine)
* No other concurrent investigational drugs
* No other concurrent cytotoxic agents
* No concurrent prophylactic fluconazole
* No concurrent or planned cyclo-oxygenase-2 (COX-2) inhibitors or nonsteroidal anti-inflammatory drugs
* No concurrent chronic use of full-dose aspirin (325 mg/day or greater)

  * Concurrent low-dose (cardioprotective) aspirin prophylaxis (no more than 325 mg every other day OR no more than 162.5 mg per day) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-05; Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus-Henning Koehne, MD, Study Chair — Klinikum Oldenburg
Locations (28):
- Belgium (6):
  - Ziekenhuis Network Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Cazk Groeninghe - Campus St-Niklaas, Kortrijk
  - St. Elizabeth Ziekenhuis, Turnhout
- National Cancer Institute - Cairo, Cairo, Egypt
- Germany (18):
  - Charite - Campus Charite Mitte, Berlin
  - General Hospital, Celle
  - Universitatsklinikum Carl Gustav Carl Carus, Dresden
  - Kliniken Essen - Mitte, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Klinikum der Albert - Ludwigs - Universitaet Freiburg, Freiburg im Breisgau
  - Allgemeines Krankenhaus Hagen, Hagen
  - Allgemeines Krankenhaus Altona, Hamburg
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - St. Marien Hospital, Hamm
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Vinzentiuskrankenhaus, Landau
  - Onkologische Schwerpunktpraxis Leer, Leer
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Kreiskrankenhaus Meissen, Meissen
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Eberhard Karls Universitaet, Tübingen
  - Universitaets-Hautklinik Wuerzburg, Würzburg
- National Institute of Oncology, Budapest, Hungary
- Israel (2):
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon

REFERENCES:
- [Result] Kohne CH, De Greve J, Hartmann JT, Lang I, Vergauwe P, Becker K, Braumann D, Joosens E, Muller L, Janssens J, Bokemeyer C, Reimer P, Link H, Spath-Schwalbe E, Wilke HJ, Bleiberg H, Van Den Brande J, Debois M, Bethe U, Van Cutsem E. Irinotecan combined with infusional 5-fluorouracil/folinic acid or capecitabine plus celecoxib or placebo in the first-line treatment of patients with metastatic colorectal cancer. EORTC study 40015. Ann Oncol. 2008 May;19(5):920-6. doi: 10.1093/annonc/mdm544. Epub 2007 Dec 6. PMID 18065406
- [Result] De Grève J, Koehne C, Hartmann J, et al.: Capecitabine plus irinotecan versus 5-FU/FA/irinotecan ± celecoxib in first line treatment of metastatic colorectal cancer (CRC). Long-term results of the prospective multicenter EORTC phase III study 40015. [Abstract] J Clin Oncol 24 (Suppl 18): A-3577, 2006.
- [Result] Kohne C, De Greve J, Bokemeyer C, et al.: Capecitabine plus irinotecan versus 5-FU/FA/irinotecan +/- celecoxib in first line treatment of metastatic colorectal cancer. Safety results of the prospective multicenter EORTC phase III study 40015. [Abstract] J Clin Oncol 23 (Suppl 16): A-3525, 252s, 2005.